CLINICAL TRIAL: NCT00494728
Title: Smoking Cessation Intervention for Depressed Smokers: Treatment Development
Brief Title: Smoking Cessation for Depressed Smokers
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0351; NCI-2012-02097 (Registry Identifier: NCI CTRP); 1R01MH076776-01A1 (NIH); 1R01MH087692 (NIH)
Record Dates: First submitted 2007-06-28; First posted 2007-07-02 (Estimated); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Smoking; Depression
Keywords: Smoking; Depression; Major Depressive Disorder; Cognitive Behavioral Analysis System of Psychotherapy; Smoking Cessation Treatment; Nicotine Replacement Therapy; Nicotine Patch; CBASP; MDD
MeSH Terms: conditions — Smoking; Depression; Depressive Disorder, Major | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CBASP + ST (Other): Cognitive Behavioral Analysis System of Psychotherapy (CBASP) + Smoking Cessation Treatment (ST)
  Interventions: Behavioral: Smoking Cessation Treatment; Drug: Nicotine Replacement Therapy; Behavioral: CBASP
- ST (Other): Smoking Cessation Treatment (ST)
  Interventions: Behavioral: Smoking Cessation Treatment; Drug: Nicotine Replacement Therapy

INTERVENTIONS:
Behavioral: Smoking Cessation Treatment — 12 60-minute individual sessions of standard smoking cessation treatment.
Drug: Nicotine Replacement Therapy — 21 mg patch for 4 weeks; 14 mg patch for 2 weeks; 7 mg patch for 2 weeks.
Behavioral: CBASP — Individual counseling sessions where taught/develop interpersonal and behavioral coping skills to help decrease depression and negative moods, and to increase ability to quit smoking.
  Other Names: Cognitive Behavioral Analysis System of Psychotherapy
  Arms: CBASP + ST

SUMMARY:
Objectives:

Primary Aim:

To conduct a preliminary randomized trial in smokers with current recurrent major depressive disorder (MDD), current MDD with a single episode of 2 years or more, and current dysthymia comparing combined cognitive behavioral analysis system of psychotherapy (CBASP) and standard smoking cessation treatment (ST) (CBASP/ST) to combined Health Education and ST treatment (HE/ST) to:

1. Examine the effects of CBASP/ST on both short and long-term point prevalence abstinence

Secondary Aims:

1. To test the hypothesis that depressed smokers in the CBASP/ST treatment will experience greater decreases in depressive symptoms from baseline to each of our follow-up assessment points, compared to depressed smokers in the HE/ST treatment, and;
2. That depressed smokers in the CBASP/ST treatment will experience greater improvements in psychosocial functioning from baseline to follow-up assessment points, compared to depressed smokers in the ST treatment.
3. To evaluate between subject neurophysiological predictors of abstinence at 3 and 6 months, and:
4. To evaluate within-subject changes in neurophysiological responses to emotional and smoking-related stimuli across treatment sessions, and the relation of these changes to abstinence and depressive symptoms at end of treatment, and 3- and 6-months.

DETAILED DESCRIPTION:
During the session today, you will be asked to complete 8-9 questionnaires about smoking history, health status, current medications you are taking, your confidence in quitting smoking, symptoms of nicotine dependence and withdrawal, symptoms of depression, negative experiences during childhood, and your thoughts and feelings about work and the quality of your relationships with others. In total, the questionnaires should take about 30-45 minutes to complete. You will also blow into a machine that measures the amount of carbon monoxide in your blood (a breath test). This visit may last 1 ½ to 2 hours.

Following the session today, you will be provided with information on the results of the screening tests you completed at BCM to see whether you have a current depressive disorder or any other psychiatric disorders. You will be provided with an opportunity to discuss this information with the investigators.

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the toss of a coin) to one of 2 groups. If you are assigned to Group 1, you will receive counseling to help develop behavioral coping skills that will help with situations where you are tempted to smoke more (which are considered high-risk situations), combined with mood management counseling to help you develop interpersonal (communication) coping skills to help with depression and negative moods that may affect your ability to quit smoking. If you are assigned to Group 2, you will receive counseling to help develop behavioral coping skills that will help with situations where you are tempted to smoke more (which are considered high-risk situations), combined with education on the health-related effects of smoking. Participants in both groups will receive nicotine patches.

During the 5 weeks after the visit, you will have six (6) 70-minute counseling sessions.

If you are in Group 1, you will receive information on how cigarette smoking is a learned habit and a physical addiction and how the habit can be unlearned. You will receive counseling to help you identify situations that are high risk for smoking and to help you develop behavioral coping plans to decrease the chances of smoking in those situations. You will be encouraged to use these skills between sessions. You will also receive counseling to help you identify situations where you interact with others that may cause negative moods. You will be taught interpersonal coping skills to help decrease depression and negative moods and to increase your ability to quit smoking and not start again. You will be given homework assignments that will help you practice these skills between sessions.

If you are in Group 2, you will receive information on how cigarette smoking is a learned habit and a physical addiction and how the habit can be unlearned. You will also receive counseling to help you identify situations that are high risk for smoking and to help you develop behavioral coping plans to decrease the chances of smoking in those situations. You will be encouraged to use these skills between sessions. You will also receive information about health issues related to smoking and you will have the opportunity to discuss this information with your counselor.

Before or after each of the counseling sessions, you will fill out 2-3 questionnaires on mood and smoking behavior and have a breath test. You will be asked to fill out 5-6 questionnaires on withdrawal symptoms, confidence in quitting smoking, your thoughts and feelings about work, and the quality of your relationships with others. In total, it will should about 30-45 minutes to fill out the questionnaires at each visit. Each of these visits will take a total of about 1 hour and 40 minutes to 1 hour and 55 minutes.

The date to quit smoking will be scheduled for about 5 weeks after your first visit. As part of your counseling sessions, you will be provided with counseling to help you develop a plan to quit and to set a quit date. You will be given the nicotine patches starting on the quit date. You will be asked to wear the nicotine patches on the upper area of your body for 24 hours each day.

Following the quit date, you will attend six (6) more 70-minute counseling sessions. You will also attend 2 additional visits at 3 months and 6 months from your quit date. At each of these visits, you will be asked to fill out 2-3 questionnaires on mood and smoking behavior and to provide a breath test to measure the amount of carbon monoxide in your blood. You will be asked questions about symptoms you may be having and the medications you are taking. You will be asked to fill out 5-6 questionnaires on withdrawal symptoms, confidence in quitting smoking, and the quality of your relationships with others at some of these visits. If you are unable to attend your end-of-treatment, 3-month or 6-month visits, you may be asked to provide a saliva sample to measure the amount of cotinine in your blood, a chemical produced by the breakdown of nicotine during smoking. This sample will be taken using a dental roll (cotton swab) placed in the mouth for several minutes to absorb saliva. At the 3-month and 6-month follow-up visits, you will be also asked questions about any current problems with depression.

At the last treatment visit (Visit 12) and at the 3-month and 6-month follow-up visits, if you are still smoking, you will be provided with information on where you can receive additional help to quit smoking. If you continue to have a current depressive disorder, you will be provided with additional information about this disorder, and you will be provided with information on where you can receive treatment for your depressive disorder. The investigators will provide a referral for treatment if you wish to receive treatment for your depressive disorder at that time.

Each of the counseling visits will be videotaped. In addition, the first visit and the visits at 3 and 6 months may also be videotaped. The videotapes will be erased within 1 year after you complete this study. The videotapes will be used to help the investigators make sure that the counselors are following the correct therapy procedures and may be used in future studies to help the investigators better understand the mood management and health education treatments. No one but the study investigators, study staff, and consultants (those who review and rate how well the study therapists follow therapy procedures) will be allowed to view the tapes. Your identity will be kept strictly confidential.

So that the study researchers can keep in contact with you throughout the study and over the long period of time between your end of treatment visit and the 3- and 6- month follow-up visits, you will be asked at the baseline visit to provide the name and address of 2 contacts (family members/friends) that you feel confident would have updated contact information on you.

Your participation in this study will end after the 6-month follow-up visit.

This is an investigational study. The nicotine patches are FDA approved for use in adults age 18 and older and commercially available. Up to 202 people will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Currently meeting DSM-IV criteria for major depressive disorder, recurrent; or major depressive disorder, recurrent, in partial remission; or major depressive disorder, single episode with a duration of 2 years or more; or; dysthymic disorder.
2. Score greater than or equal to 8 on the PHQ at baseline
3. Age greater than or equal to 16
4. Smoking greater than or equal to 5 cigarettes per day
5. Willing to set a quit date within 6 weeks of baseline
6. English speaking and have a telephone
7. Willing to attend all sessions
8. Willing to provide informed consent and agree to all assessments and study procedures

Exclusion Criteria:

1. History of psychotic or bipolar disorder
2. Current psychotherapy
3. Current use of antidepressant
4. Current principal DSM-IV Axis I disorder other than unipolar depression or nicotine dependence
5. Involvement in any smoking cessation activities
6. Current use of nicotine replacement therapy
7. Known health or other complications that would adversely affect attendance
8. Severe levels of depressive symptoms, vegetative symptoms, and/or symptoms related to secondary psychiatric disorders that place participant at risk for harm or require immediate treatment
9. Currently at severe or extreme risk of suicide or moderate risk with resolved plans and preparation
10. Medical contraindications for use of nicotine patch, including uncontrolled heart disease, history of severe hypersensitivity to nicotine replacement products, or currently pregnant or lactating
11. 11) History of current medical condition, or any other factor that, in the judgment of the principal investigator, would likely preclude completion of study requirements.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2007-06-28 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Abstinence Rates | Approximately each 12 weeks following end of treatment (about 6 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Blalock, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org